CLINICAL TRIAL: NCT06688734
Title: Suction Versus Water Seal for Initial Treatment of Traumatic Pneumothorax Trial
Acronym: SEAL IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Eric Yeates, Acute Care surgery Clinical Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 241132
Record Dates: First submitted 2024-11-10; First posted 2024-11-14 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Pneumothorax; Trauma
Keywords: traumatic; trauma; pneumothorax; chest tube; duration
MeSH Terms: conditions — Pneumothorax; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Alternating each month, patients with traumatic pneumothoraces receiving chest tubes will have their chest tubes placed to either water seal or suction initially. The remainder of the chest tube management will be left to the provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Initial Water Seal (Experimental): After chest tube placement, the chest tube will be placed to 20cm H2O of suction for 1 minute to evacuate all pneumothorax. After this, the chest tube will be placed to water seal, defined as the water seal chamber on the chest tube drainage system being filled up to the 2cm line and not on suction. All other management decisions related to the chest tube will be left to the providers.
  Interventions: Procedure: Inital water seal
- Initial Suction (Experimental): After chest tube placement, the suction group will have their chest tube placed to 20cm H2O of suction delivered by the chest tube drainage suction. All other management decisions related to the chest tube will be left to the providers.
  Interventions: Procedure: Initial suction

INTERVENTIONS:
Procedure: Inital water seal — After chest tube placement, the chest tube will be placed to 20cm H2O of suction for 1 minute to evacuate all pneumothorax. After this, the chest tube will be placed to water seal, defined as the water seal chamber on the chest tube drainage system being filled up to the 2cm line and not on suction. All other management decisions related to the chest tube will be left to the providers.
  Arms: Initial Water Seal
Procedure: Initial suction — After chest tube placement, the suction group will have their chest tube placed to 20cm H2O of suction delivered by the chest tube drainage suction. All other management decisions related to the chest tube will be left to the providers.
  Arms: Initial Suction

SUMMARY:
The goal of this clinical trial is to compare the effect of placing chest tubes to water seal versus suction initially, in patients with traumatic pneumothoraces, on overall chest tube duration.

The main question it aims to answer is:

* Does placing chest tubes to water seal initially results in a shorter chest tube duration, without an increase in complications?

Alternating each month, patients' chest tubes will either be placed to water seal or to suction initially. All other management decisions related to the chest tube will be left to the providers.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the trauma surgery service
* pneumothorax requiring a chest tube

Exclusion Criteria:

* less than 18 years olf
* pregnant
* prisoner
* greater than 300cc of hemothorax on CT
* chest tube placed prior to CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Chest tube duration | Through study completion, an average of 1 year
  Duration of the initial chest tube, measured in hours

SECONDARY OUTCOMES:
Change from water seal to suction | Through study completion, an average of 1 year
  Yes/No
Additional chest tube placement on affected side | Through study completion, an average of 1 year
  Yes/no
Pneumothorax reaccumulation with chest tube to water seal | Through study completion, an average of 1 year
  Yes/no Yes if growth of pneumothorax on chest x-ray with tube to water seal
Replacement of chest tube | Through study completion, an average of 1 year
  Yes/no Yes if chest tube removed and then a new one is place on the same side at a later time
Pneumothorax reaccumulation after chest tube removal | Through study completion, an average of 1 year
  Yes/no Yes if pneumothorax grows on chest x-ray after chest tube removal
Hypoxic events | Through study completion, an average of 1 year
  Yes/no Yes if <90% O2 saturation is recorded in chart
Empyema | Through study completion, an average of 1 year
  Yes/no Yes if clinically diagnosed by provider based off of imaging, operative findings, clinical picture, culture results, or operative findings
Pneumonia | Through study completion, an average of 1 year
  Yes/no Yes if clinically diagnosed and treated for pneumonia
Retained hemothorax | Through study completion, an average of 1 year
  Yes/no Yes if >300cc hemothorax seen on CT scan after chest tube placement
TPA administration | Through study completion, an average of 1 year
  Yes/no Yes if any TPA administered to the affected side of the chest
Chest tube site, skin and soft tissue infection | Through study completion, an average of 1 year
  Yes/no Yes if skin and soft tissue infection treated with incision and drainage, or antibiotics
Video-assisted thoracoscopic surgery | Through study completion, an average of 1 year
  Yes/no Yes if receives video-assisted thoracoscopic surgery on the affected side during initial admission
Acute respiratory failure requiring intubation | Through study completion, an average of 1 year
  Yes/no Yes if intubated for hypoxia or hypercapnea during hospital stay
Unplanned ICU admission | Through study completion, an average of 1 year
  Yes/no Yes if admitted to ICU unexpectedly, for clinical deterioration
30-day mortality | Through study completion, an average of 1 year
  Yes/no Yes if died within 30 days of initial presentation
Length of hospital stay | Through study completion, an average of 1 year
  Integer, measured in days, length of initial hospital stay
30-day readmission | Through study completion, an average of 1 year
  Yes/no Yes if readmitted within 30 days of discharge
Thoracic intervention during readmission | Through study completion, an average of 1 year
  Yes/no Yes if readmitted and receives chest tube, video-assisted thoracoscopic surgery, or thoracotomy on the affected side

OTHER OUTCOMES:
Size of residual pneumothorax on first chest x-ray | Through study completion, an average of 1 year
  Measured in cm, largest distance from lung edges to chest wall
Presence of air leak each day | Through study completion, an average of 1 year
  Yes/no Recorded each day there is a chest tube present
Number of chest x-rays | Through study completion, an average of 1 year
  Integer, number of chest x-rays after initial trauma evaluation
Number of CT scans of chest after initial imaging | Through study completion, an average of 1 year
  Integer value Number of CT scans of chest after initial trauma evaluation during hospital stay
Chest tube related costs | Through study completion, an average of 1 year
  Integer, dollar amount Total cost of chest tube supplies utilized, imaging (chest x-rays plus CT scans of chest), operative room costs if applicable, hospital days
Mechanical ventilation | Through study completion, an average of 1 year
  Yes/no Yes if was on mechanical ventilation at any point during hospitalization
Length of ICU stay | Through study completion, an average of 1 year
  Total times spent in the ICU, measured in days
Discharge disposition | Through study completion, an average of 1 year
  Categorical Home, inpatient rehab, skilled nursing facility, long term acute care hospital, or died

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feenstra TM, Dickhoff C, Deunk J. Systematic review and meta-analysis of tube thoracostomy following traumatic chest injury; suction versus water seal. Eur J Trauma Emerg Surg. 2018 Dec;44(6):819-827. doi: 10.1007/s00068-018-0942-7. Epub 2018 Mar 15. PMID 29546613
- [Background] Muslim M, Bilal A, Salim M, Khan MA, Baseer A, Ahmed M. Tube thorocostomy: management and outcome in patients with penetrating chest trauma. J Ayub Med Coll Abbottabad. 2008 Oct-Dec;20(4):108-11. PMID 19999219
- [Background] Majumdar MNI, et al. Role of Continuous low pressure suction in management of traumatic haemothorax and/or haemopneumothorax: experiences at NIDCH and CMH Dhaka. J Armed Forces Med Coll (JAFMC) Bangladesh. 2014;10(2):21-26.
- [Background] Morales CH, Mejia C, Roldan LA, Saldarriaga MF, Duque AF. Negative pleural suction in thoracic trauma patients: A randomized controlled trial. J Trauma Acute Care Surg. 2014 Aug;77(2):251-5. doi: 10.1097/TA.0000000000000281. PMID 25058250
- [Background] Marshall MB, Deeb ME, Bleier JI, Kucharczuk JC, Friedberg JS, Kaiser LR, Shrager JB. Suction vs water seal after pulmonary resection: a randomized prospective study. Chest. 2002 Mar;121(3):831-5. doi: 10.1378/chest.121.3.831. PMID 11888968
- [Background] Cerfolio RJ, Bass C, Katholi CR. Prospective randomized trial compares suction versus water seal for air leaks. Ann Thorac Surg. 2001 May;71(5):1613-7. doi: 10.1016/s0003-4975(01)02474-2. PMID 11383809
- [Background] Anderson D, Chen SA, Godoy LA, Brown LM, Cooke DT. Comprehensive Review of Chest Tube Management: A Review. JAMA Surg. 2022 Mar 1;157(3):269-274. doi: 10.1001/jamasurg.2021.7050. PMID 35080596
- [Background] Di Bartolomeo S, Sanson G, Nardi G, Scian F, Michelutto V, Lattuada L. A population-based study on pneumothorax in severely traumatized patients. J Trauma. 2001 Oct;51(4):677-82. doi: 10.1097/00005373-200110000-00009. PMID 11586158